CLINICAL TRIAL: NCT04991545
Title: Feasibility of the RetrogradeTranscutaneous Infra-Red Illumination for Facilitation of Video Scope-tracheal Intubation
Brief Title: Feasibility of the Infra-Red Illumination for Facilitation of Video Scope-tracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MRC-05-088
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Airway Morbidity; Covid19; Trachea
Keywords: Infra-Red Illumination; Retrograde Transcutaneous; videoscope-tracheal Intubation
MeSH Terms: conditions — COVID-19; Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: control group (intubation without IRD/IRRIS device) (No Intervention): Group A = control group (intubation without IRD/IRRIS device) (15 subjects) The first operator experienced with video-laryngoscopy intubation will do the endotracheal intubation after induction of anesthesia.
- Intervention group using Infrared (Active IRD/ IRRIS) device (Experimental): Group B = intervention group using Infrared active IRD/IRRIS device (15 subjects) Before inducing anesthesia, the second operator will open the randomization envelope and adhere IRRIS/IRD device to the anterior skin of the neck above the sternal notch according to the group of patients. After confirming lack of discomfort during application of the IRRIS/IRD device, anesthesia will be induced
  Interventions: Device: Application of Infrared (Active IRD/ IRRIS) device

INTERVENTIONS:
Device: Application of Infrared (Active IRD/ IRRIS) device — The first operator experienced with video-laryngoscopy intubation will do Before inducing anesthesia, the second operator will open the randomization envelope and adhere IRRIS/IRD device to the anterior skin of the neck above the sternal notch according to the group of patients After confirming lack of discomfort during application of the IRRIS/IRD device,
  After complete relaxation, Laryngoscopy will be performed by the first operator using video laryngoscope (Glidescope Verathon Medical, BC, Canada or C-Mac Storz, Germany) to insert the tracheal tube. The endotracheal tube will be armed with a malleable stylet and to be molded to a curved 'hockey stick or the same curve of the laryngoscopic blade's shape. We will divide the patient according to device into two groups:
  1. Group A: control group
  2. Group B: Intervention group using Infrared
  Arms: Intervention group using Infrared (Active IRD/ IRRIS) device

SUMMARY:
Airway securing through the placement of an endotracheal tube continues to be the definitive and the global standard management. The successful first attempt is aimed to avoid the consequences of multiple intubation trials as bleeding, tissue swelling, and airway contamination from gastric content that led to considerable morbidity and mortality. Visualization of the larynx and the glottic opening is the key to first-pass success requiring long-term training and availability of specific equipment concerned to that. For confirmation of the position endotracheal tube or its displacement, various clinical and equipment aids to that which are not valid or limited in different scenarios. Video laryngoscopes (VL) have been proposed to improve laryngeal visualization, hence a higher first-pass success rate accomplished. Despite that, there are limitations of video laryngoscope use in different circumstances that requiring adding of other aids to facilitate endotracheal intubation.

x

DETAILED DESCRIPTION:
Airway securing through the placement of an endotracheal tube continues to be the definitive and the global standard management. The successful first attempt is aimed to avoid the consequences of multiple intubation trials as bleeding, tissue swelling, and airway contamination from gastric content that led to considerable morbidity and mortality. Visualization of the larynx and the glottic opening is the key to first-pass success requiring long-term training and availability of specific equipment concerned to that. For confirmation of the position endotracheal tube or its displacement, various clinical and equipment aids to that which are not valid or limited in different scenarios. Video laryngoscopes (VL) have been proposed to improve laryngeal visualization, hence a higher first-pass success rate accomplished. Despite that, there are limitations of video laryngoscope use in different circumstances that requiring adding of other aids to facilitate endotracheal intubation.

The proposal of this study is to assess the feasibility and the impact of infrared/near-infrared (IRD) light on the performance of video-laryngoscopy and reduction of the time needed for endotracheal intubation and increase the credibility of the device.

Data-collection will be started after induction of the anesthesia and ended at the confirmation of endotracheal tube position

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* General anesthesia that needs endotracheal intubation
* All Mallampati score 1-3
* ASA physical status 1-3

Exclusion Criteria:

* Refuse or unable to sign the consent.
* Pregnancy
* Emergency cases
* History of or expected difficult intubation
* Maxillofacial abnormality or trauma
* Age below 18 years
* Rapid sequence induction
* Skin disorders and skin light sensitivity (SLE, Lupus ….)
* Impaired head and neck mobility
* Scars or skin injuries at the neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
infrared red light on the performance of video-laryngoscopy intubation and its impact on first pass success | During procedure time
  The primary endpoint will be the feasibility of infrared/near-red light on the performance of video-laryngoscopy tracheal intubation and its impact on first pass success

SECONDARY OUTCOMES:
Visibility of the glottic entrance | During procedure time
  Visibility of the glottic entrance during intubation
Time to recognize the illuminated laryngeal inlet. | one year
  Time to recognize the illuminated laryngeal inlet.
Correct intubation | one year
  Recognize the correct intubation pathway by other confirmatory tests
Number of intubation attempt. | During procedure time
  Number of intubation attempt by the experience staff.
Types of video laryngoscopy | During procedure time
  Types of video laryngoscopy used
Alternative techniques of intubation. | During procedure time
  Alternative techniques of intubation if used after failure of primary equipment
Safety of Infra Red | During procedure time
  Safety: Presence and severity of skin lesion that might be associated at device application site. (Discomfort, pressure sign, irritation, redness, burn)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Shallik, M.D., Principal Investigator — Hamad Medical Corporation - HMC
Locations (1):
- ACC&HGH, Hamad Medical Corporation, Doha, Doah, Qatar

IPD SHARING:
Plan to Share IPD: Yes
We will share the data after IRB approval
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After IRB approval directly
Access Criteria: Website

REFERENCES:
- [Result] Simpson GD, Ross MJ, McKeown DW, Ray DC. Tracheal intubation in the critically ill: a multi-centre national study of practice and complications. Br J Anaesth. 2012 May;108(5):792-9. doi: 10.1093/bja/aer504. Epub 2012 Feb 6. PMID 22315326
- [Result] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Result] Webb RK, Currie M, Morgan CA, Williamson JA, Mackay P, Russell WJ, Runciman WB. The Australian Incident Monitoring Study: an analysis of 2000 incident reports. Anaesth Intensive Care. 1993 Oct;21(5):520-8. doi: 10.1177/0310057X9302100507. PMID 8273871
- [Result] Duggan LV, Mastoras G, Bryson GL. Tracheal intubation in patients with COVID-19. CMAJ. 2020 Jun 1;192(22):E607. doi: 10.1503/cmaj.200650. Epub 2020 May 1. No abstract available. PMID 32357995
- [Result] Knapp S, Kofler J, Stoiser B, Thalhammer F, Burgmann H, Posch M, Hofbauer R, Stanzel M, Frass M. The assessment of four different methods to verify tracheal tube placement in the critical care setting. Anesth Analg. 1999 Apr;88(4):766-70. doi: 10.1097/00000539-199904000-00016. PMID 10195521
- [Result] Nemec D, Austin PN, Silvestro LS. Methods to Improve Success With the GlideScope Video Laryngoscope. AANA J. 2015 Dec;83(6):389-97. PMID 26742332
- [Result] Saima S, Asai T, Kimura R, Terada S, Arai T, Okuda Y. [Combined Use of a Videolaryngoscope and a Transilluminating Device for Intubation with Two Difficult Airways]. Masui. 2015 Oct;64(10):1045-7. Japanese. PMID 26742405
- [Result] Kristensen MS, Fried E, Biro P. Infrared Red Intubation System (IRRIS) guided flexile videoscope assisted difficult airway management. Acta Anaesthesiol Scand. 2018 Jan;62(1):19-25. doi: 10.1111/aas.13016. Epub 2017 Oct 24. PMID 29063583
- [Result] Wayne MA, McDonnell M. Comparison of traditional versus video laryngoscopy in out-of-hospital tracheal intubation. Prehosp Emerg Care. 2010 Apr-Jun;14(2):278-82. doi: 10.3109/10903120903537189. PMID 20199237